CLINICAL TRIAL: NCT05799846
Title: Adapting Episodic Future Thinking for Behavioral Weight Loss: Comparing Strategies and Characterizing Treatment Response
Brief Title: Cognitive Strategies for Weight Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Brown University (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Kathryn E. Demos, Asst. Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1809657-4; R01DK128412 (NIH)
Record Dates: First submitted 2023-02-28; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STANDARD Behavioral (Active Comparator): This is a 12-month Internet-delivered behavioral weight loss (iBWL) program that has been used in numerous studies and is currently considered our 'standard' treatment. Participants are asked to adhere to calorie and physical activity (PA) goals and are required to self-monitor weight, intake, and PA daily via a study website. Participants will have a training session prior to beginning iBWL to learn about the website and their specific weight-related goals. The iBWL includes 3 months of weekly video lessons teaching skills to modify eating and PA behaviors. These lessons and individualized feedback to participants incorporate key BWL strategies. Participants will then have a 'refresher' training session at 3 months to discuss standard behavioral weight loss strategies and help control for contact across arms. For the remainder of the program (months 4-12) participants will have monthly lessons, self-monitoring (tracking calories and PA 1 wk/month) and feedback.
  Interventions: Behavioral: Standard Behavioral Weight Loss Intervention
- PREVENT (Experimental): This is a 12-month Internet-delivered behavioral weight loss (iBWL) program in which participants are asked to adhere to calorie and physical activity (PA) goals and are required to self-monitor weight, intake, and PA daily via a study website. Additionally, PREVENT uses a future-oriented cognitive strategy featuring Episodic Future Thinking (EFT) to focus on long-term negative consequences of unhealthy choices. Participants will receive training in PREVENT strategies prior to beginning iBWL. The iBWL includes 3 months of weekly video lessons teaching skills to modify eating and PA behaviors. These lessons and individualized feedback to participants are framed according to PREVENT (i.e., focusing on avoiding long-term consequences of unhealthy choices) and include specific exercises and reminders to use the strategy. Participants will then have a 'refresher' training session at 3 months, followed by monthly lessons, self-monitoring (tracking calories and PA 1 wk/month) and feedback.
  Interventions: Behavioral: PREVENT Behavioral Weight Loss Intervention
- PROMOTE (Experimental): This is a 12-month Internet-delivered behavioral weight loss (iBWL) program in which participants are asked to adhere to calorie and physical activity (PA) goals and are required to self-monitor weight, intake, and activity daily via a study website. Additionally, PROMOTE uses a future-oriented cognitive strategy featuring Episodic Future Thinking (EFT) to focus on long-term benefits of healthy choices. Participants will receive cognitive training in PROMOTE prior to beginning iBWL. The iBWL includes 3 months of weekly video lessons teaching skills to modify eating and activity behaviors. These lessons and individualized feedback to participants are framed according to PROMOTE (i.e., focusing on achieving long-term benefits of healthy choices) and include specific exercises and reminders to use the strategy. Participants will then have a 'refresher' training at 3 months, followed by monthly lessons, self-monitoring (tracking calories and PA 1 wk/month), and feedback.
  Interventions: Behavioral: PROMOTE Behavioral Weight Loss Intervention

INTERVENTIONS:
Behavioral: Standard Behavioral Weight Loss Intervention — 12-month online behavioral weight loss intervention
  Arms: STANDARD Behavioral
Behavioral: PREVENT Behavioral Weight Loss Intervention — 12-month online behavioral weight loss intervention focused on preventing future negative consequences of obesity
  Arms: PREVENT
Behavioral: PROMOTE Behavioral Weight Loss Intervention — 12-month online behavioral weight loss intervention focused on promoting future benefits of maintaining a healthy weight
  Arms: PROMOTE

SUMMARY:
The goal of this clinical trial is to compare weight change and other related outcomes associated with three different behavioral weight loss interventions (STANDARD Behavioral, PREVENT, and PROMOTE) in adults with obesity. The main questions it aims to answer are:

* Which of the three Internet-delivered weight loss programs results in the greatest weight loss?
* How do key weight-related behaviors (e.g., adherence, diet, physical activity) differ across the arms?
* What individual characteristics predict success in each arm?
* What are the underlying mechanisms of each approach?
* Are there any potential adverse outcomes associated with any of the conditions (e.g., depression, weight stigmatization, increased body image concerns).

Participants will:

* signed informed consent
* complete a baseline assessment
* be randomized to 12 months of either Standard iBWL, PREVENT or PROMOTE
* complete a training workshop to learn arm-specific cognitive strategies
* complete a 12-month Internet-delivered weight loss program, requiring self-monitoring of intake and exercise and viewing of 12 weekly lessons followed by 9 monthly lessons
* complete an assessment at 3 months (during treatment)
* complete a refresher workshop on arm-specific cognitive strategies at 3 months
* complete an assessment at 6 months (during treatment), 12 months (at the conclusion of treatment), and 18 months (6 months after treatment

ELIGIBILITY:
Inclusion Criteria:

* Participants will be between the ages of 18 and 70, have a BMI between 25 and 45 kg/m2, and have regular (i.e., weekly) access to the Internet, defined as owning a smart phone with Internet capabilities, and/or having a broadband or Wi-Fi connection at home or work.

Exclusion Criteria:

* Exclusionary criteria include: 1) current enrollment in a weight loss program, 2) currently taking weight loss medications, 3) history of bariatric surgery or planned bariatric surgery in the next 18 months, 4) individuals who are pregnant, nursing, or have plans to become pregnant within the next 18 months, 5) individuals planning to relocate outside the area in the next 18 months, 6) any medical condition for which weight loss would be contraindicated, 7) neurological or psychiatric conditions including but not limited to schizophrenia and bipolar disorder, 8) inability to attend assessments at the Weight Control and Diabetes Research Center in Providence, RI.

Individuals with mobility issues, dizziness, or history of heart disease, diabetes, or cancer will be required to provide physician consent prior to enrolling.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Percent Weight Change at 3 months | 3 months after randomization
  Weight change is the primary outcome in this trial and will be calculated as change from baseline.
Percent Weight Change at 6 months | 6 months after randomization
  Weight change is the primary outcome in this trial and will be calculated as change from baseline.
Percent Weight Change at 12 months | 12 months after randomization
  Weight change is the primary outcome in this trial and will be calculated as change from baseline.
Percent Weight Change Post-Treatment | 18 months after randomization
  Post-treatment weight change will be calculated as percent weight change observed at the 18 month assessment (6 months following treatment completion)

SECONDARY OUTCOMES:
Change in Actigraph-measured Physical Activity (PA) | 12 months after randomization
  To address Secondary Aim 1, physical activity (PA) will be objectively-measured for 1 week at baseline, 3m, 12m, and 18m using ActigraphGT9X Link. Participants will be instructed to wear the accelerometer on their waist during all waking hours, exclusive of bathing and swimming, for 7 consecutive days. This monitor uses a validated triaxial accelerometer and proprietary data filtering technology to estimate free-living PA and sedentary behaviors. Accelerometer data will be processed and analyzed using Actigraph's ActiLife software. Data will be considered valid if the monitor was worn for more than 10 hours on more than 4 days (including one or more weekend day). Intensity will be assessed as average counts per minute (cpm) and previously validated cut points (Freedson et al., 1998) will be used to identify bout-related moderate-to-vigorous intensity PA (greater than or equal to 1952 cpm accumulated in bouts greater than or equal to 10 min) and sedentary time (less than 100 cpm).
Change in Dietary Recall | 12 months after randomization
  Diet will be measured through 3, non-consecutive 24-hour diet recalls at baseline, 3m, 12m, and 18m. Recalls will be collected on two weekdays and one weekend at each time point with the first recall collected during the in-person assessment and the subsequent two recalls collected via phone. A trained interviewer will collect recalls using Nutrition Data Systems for Research (NDSR 2018; Nutrition Coordinating Center, University of Minnesota). NDSR uses a multipass method which provides participants multiple opportunities to recall each consumed food/beverage and reduces reporting biases. Given issues with use of dietary recalls to determine absolute energy intake, NDSR output will be used to examine changes in energy density and diet quality, as measured by the Healthy Eating Index, 2015 (HEI-2015). Component scores will highlight changes in intake of fruits and vegetables, whole grains, and lean proteins as well as calories from alcohol, added sugars and energy-dense snacks.
Intervention Adherence - lessons viewed | 12 months after randomization
  Intervention adherence will be assessed automatically via the study website during the entire 12-month iBWL treatment program. Outcome measures will include number of website number of intervention videos viewed.
Intervention Adherence - self-monitoring | 12 months after randomization
  Intervention adherence will be assessed automatically via the study website during the entire 12-month iBWL treatment program. Outcome measures will include number of website number of self-monitoring entries during the weight loss program.

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control & Diabetes Research Center, Providence, Rhode Island, United States